CLINICAL TRIAL: NCT06235528
Title: A Cross Sectional Prospective Study on Critically Ill Children Admitted in PICU of Children's Hospital Assuit University
Brief Title: Gastrointestinal Manifestations in Critically Ill Children Admitted in PICU of Children's Hospital Assuit University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abdalla Hashem Ahmed, 71515, Assuit University, Assiut University
Other Study IDs: GIT manifestations
Record Dates: First submitted 2023-12-09; First posted 2024-02-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Gastrointestinal Manifestations in Critically Ill Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal complications are common in critically ill children. GIC are commonly observed, as either a primary reason for admission or as a part of multiple organ dysfunction syndromes MODS in children admitted in the Pediatric Intensive Care Unit (PICU). Despite its prominence in critically ill patients with MODS.

GIC are often ignored in PICU which often delays enteral nutrition preventing patients from getting adequate calorie and protein intake, ultimately leading to acquired malnutrition in these patients. The lack of a uniform standard definition of GIC adds to delays in its recognition. Critical illness can result in intestinal mucosal ischemia that further damages the gut barrier function

DETAILED DESCRIPTION:
Gastrointestinal complications are common in critically ill children. GIC are commonly observed, as either a primary reason for admission or as a part of multiple organ dysfunction syndromes in children admitted in the Pediatric Intensive Care Unit . Despite its prominence in critically ill patients with MODS.

GIC are often ignored in PICU which often delays enteral nutrition preventing patients from getting adequate calorie and protein intake, ultimately leading to acquired malnutrition in these patients. The lack of a uniform standard definition of GIC adds to delays in its recognition. Critical illness can result in intestinal mucosal ischemia that further damages the gut barrier function.

Recently with the increasing awareness of GIC in critically ill patients, the Working Group on Abdominal Problems of the European Society of Intensive Care Medicine proposed a set of definitions of acute gastrointestinal injury in critical illnesses in adults for both clinical and research purposes. However, there is no such definition available for the pediatric population. Also, the associations between AGI grades, the severity of GI dysfunction and adverse outcome remains to be elucidated.

Reintam et al reported an incidence of GIC of 59% in their mixed-ICU population. Common GIC included vomiting, high gastric residual volume , bowel distension, diarrhea, and GI bleeding, in their report. There is limited published literature on the frequency and outcome of GIC related to enteral feeding in critically ill children. Critically ill patients with GIC have a prolonged length of stay in ICU and higher mortality as compared to those without Gastrointestinal complications The most common symptoms of GIT issues, regardless of cause, are vomiting and diarrhea. Gastroenteritis resulting from an infection can also cause fever. Abdominal pain is also common.

Most encountered gastrointestinal problems in critically ill children will be discussed:

•Dehydration, Gastrointestinal bleeding, Dysmotility, Constipation, Malnutrition

1. Dehydration:

   The most common cause of dehydration in young children is severe diarrhea and vomiting. Older adults naturally have a lower volume of water in their bodies, and may have conditions or take medications that increase the risk of dehydration.

   , seriously dehydrated children become listless, irritable, or sluggish . Infants are much more likely than older children to become dehydrated and develop serious side effects. Infants who are dehydrated need medical care right away.
2. Gastrointestinal Bleeding:

   GI bleeding is associated with risk factors such as respiratory failure, coagulopathy, or PRISM score >10.

   Pathophysiology is complex and begins with vasoconstriction and ischemia, eventually leading to bleeding that results from stress ulcerations, called stress ulcer-related bleeding . Upper GI bleeding has different pathophysiological mechanisms, for example, in acid reflux-related esophagitis. It has also been documented that acid suppression does not prevent UGIB or SURB. Stress ulcers are caused by decreased mucosal blood flow and reperfusion injury and less related to chronic acid secretion-related peptic ulcers. Exact pathophysiology is not fully understood.
3. Dysmotility In the critically ill child causes delayed gastric emptying (GE) or gastroparesis. It has been reported in up to 50% of critically ill children. Potential for aspiration, ventilator-associated pneumonia, inadequate enteral nutrition, and resulting poor efficacy of enteral medications results in poor patient outcomes.

   Gastric dysmotility in a critically ill child may accompany gastroesophageal reflux , with high risk for aspiration and ventilator-associated pneumonia in mechanically ventilated patients.
4. Constipation Constipation in a critically ill child is a poorly studied disease which can represent up to 50% of children admitted to Pediatric Intensive Care Units.

   In one pediatric study, it was found to be common in postsurgical, older, and obese children and ones with fecal continence p value < 0.01. Patients with constipation had higher severity PIM2: Pediatric Index of Mortality 2 scores and started nutrition later and with a lower volume p value < 0.01. Overall management included enemas and/or oral laxatives. Major independent risk factors are body weight, PIM2 clinical severity score, ICU admission after surgery, and the need for vasoconstrictor therapy, resulting in intestinal hyperpermeability as well as associated therapies such as vasoconstrictor therapy, and overall management mainly remains empirical.
5. Malnutrition In the ill child, malnutrition is usually of multifactorial origin. It is associated with an altered metabolism of certain substrates, increased or decreased metabolism and catabolism depending on the severity and kind of the lesion, and reduced nutrient delivery. The presence of malnutrition prior to admission worsens the prognosis in the critically ill child and, furthermore, severe illness has marked repercussions on the nutritional status of these patients Malnutrition interferes with the appropriate response of the body to disease and predisposes to infection and to the onset of multiorgan failure, increasing morbidity and mortality, the mean length of hospital stay, and health costs.

ELIGIBILITY:
Inclusion criteria

• All children admitted to PICU with age one month to 18 years of both gender and have developed GIT manifestations after admission as a sequel of other diseases (intestinal perforation, intestinal obstruction, necrotizing fasciitis…)

Exclusion Criteria:

* Age more than 18 years old
* Children have no GIT Complications

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children admitted to PICU who have GIT manifestations after admission as sequel of other diseases
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
describe demographic and clinical data of critically ill children with Gastrointestinal manifestations admitted to PIUC | 2 years
  Describe the distribution of etiologies of Gastrointestinal manifestations admitted to PIUC,The most common symptoms of GIT issues, regardless of cause, are vomiting and diarrhea. Gastroenteritis resulting from an infection can also cause fever. Abdominal pain is also common